CLINICAL TRIAL: NCT03640403
Title: Effectiveness and Safety of Intermittent Preventive Treatment for Malaria Using Either Dihydroartemisinin-piperaquine or Artesunate-amodiaquine in Reducing Malaria Related Morbidities and Improving Cognitive Ability in School-aged Children in Tanzania: A Controlled Randomised Trial
Brief Title: Effectiveness and Safety of Intermittent Preventive Treatment for Malaria Using Either Dihydroartemisinin-piperaquine or Artesunate-amodiaquine in Reducing Malaria Related Morbidities and Improving Cognitive Ability in School-aged Children in Tanzania
Acronym: InSMART-school
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute for Medical Research, Tanzania (Other Government)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Dr. Geofrey Makenga, Principal Investigator, National Institute for Medical Research, Tanzania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TEAM VERSION3
Record Dates: First submitted 2018-08-14; First posted 2018-08-21 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Malaria,Falciparum; Anemia
Keywords: Malaria; school children; randomized controlled trial; safety; effectiveness; Dihydroartemisinin-piperaquine; cognitive; Artesunate-amodiaquine; malaria serology; drug resistance
MeSH Terms: conditions — Malaria, Falciparum; Anemia; Malaria | interventions — amodiaquine, artesunate drug combination

STUDY DESIGN:
Intervention Model Description: A randomized, controlled, open label study assessing the effectiveness and safety of 2 antimalarial drugs for IPTsc, namely DP and ASAQ by a 3-arm trial using a "balanced block design" with the "standard of care" arm as reference.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DP (Experimental): Dihydroartemisinin-piperaquine (DP), antimalarial drug to be given every 4 months 3 rounds for the first year. A second non-interventional year will assess possible rebound effects.
  Interventions: Drug: Dihydroartemisinin-piperaquine
- ASAQ (Active Comparator): Artesunate-amodiaquine (ASAQ), antimalarial drugs to be given every 4 months 3 rounds for the first year. A second non-interventional year will assess possible rebound effects.
  Interventions: Drug: Artesunate-amodiaquine
- Control (No Intervention): No intervention drugs will be given, but normal routine standard of care will be provided.

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine — Dihydroartemisinin-piperaquine (DP). One of the Artemisinin combination therapy(ACTs), indicated for treatment of uncomplicated malaria. It will to be given every 4 months 3 rounds for a year.
  Arms: DP
Drug: Artesunate-amodiaquine — Artesunate-amodiaquine (ASAQ). One of the Artemisinin combination therapy(ACTs), indicated for treatment of uncomplicated malaria. It will to be given every 4 months 3 rounds for a year.
  Arms: ASAQ

SUMMARY:
Background:

In high-transmission settings, up to 70% of school-aged children harbour malaria parasites which is mostly asymptomatic, thus, from an epidemiological point of view, they contribute significantly as reservoir to onward malaria transmission to others. In endemic areas, malaria accounts for around 50% of the mortality, 13-50% of all school absenteeism, and causes anaemia in approximately 85 million school-aged children of sub Saharan Africa that also impairs the cognitive development of children. Intermittent preventive treatment (IPT) of pregnant women as well as seasonal malaria chemoprevention in children under the age of five have been implemented in several sub-Saharan countries and have proven to be very effective. However, none of these IPT strategies is targeting school children. A clinical trial is being conducted to expand the IPT by testing effectiveness and safety of two antimalarial drugs Dihydroartemisinin-piperaquine (DP) and Artesunate-amodiaquine (ASAQ) in preventing malaria related morbidity in school aged children (IPTsc) living in high endemic areas.

Methods:

A randomized, open label, controlled trial will enrol 1602 school children aged 5-15 years, who will receive either DP or ASAQ or control (no drug ), using a "balanced block design" with the "standard of care" arm as reference. The interventional treatments are given every 4 months 3 rounds for the first year. A second non-interventional year will assess possible rebound effects. All study-arms receive bed nets, early diagnosis and care for malaria, and praziquantel and albendazole as mass treatment for helminthiasis. The primary endpoint are change from baseline in mean haemoglobin concentration at months 12 and 20 of follow-up and clinical malaria incidence from month 0 till months 12 and 20 of follow up. Adverse events will be monitored throughout the study. Mixed design methods will be used to assess the acceptability, cost-effectiveness and feasibility of this IPTsc as part of a more comprehensive school children health package.

Discussion:

The national school health programme (NSHP), Tanzania, combines schistosomiasis and soil transmitted helminthes (STH) control package under national schistosomiasis and STH control programme (NSSCP). Malaria intervention using IPTsc strategy may be integrated in NSHP with the same platform as NSSCP, however, there is limited systematic evidence to assess the operational feasibility of this approach. School aged children are a reachable target population in any endemic malaria setting. The suggested strategy will provide effective protection against malaria, hasten either the elimination process and/or diminish the reservoir and burden.

ELIGIBILITY:
Inclusion Criteria:

* Includes parental/guardian informed consent
* Assent by primary school children aged 11 years and above.
* Aged 5-15 years.
* Currently, lives within the pre-defined catchment area of Muheza District.
* Will remain within the same area throughout the study period (preferably class five and below).

Exclusion Criteria:

* Students at class 6 and 7
* Currently enrolled in another study or participated in another investigational drug study within the last 30 days.
* Known to have heart disease or a known cardiac ailment.
* Reports known hypersensitivity to the study drugs.
* Not willing to undergo all study procedures including physical examination and to provide blood samples as per this study protocol.
* Having clinical features of severe anaemia
* Febrile due to non-malaria illness at the time of recruitment.
* Has apparent severe infection or any condition that requires hospitalization
* Illness or conditions like hematologic, cardiac, renal, hepatic diseases which in the judgement of the investigator would place the subject at undue risk or interfere with the results of the study, including known G6PD deficiency and SS sickle cell.
* Body weight < 14 k

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1555 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean haemoglobin concentration at months 12 and 20 of follow-up | at months 0, 12 and 20
  Will measure change from baseline haemoglobin concentration at month 12 (intervention period) and at month 20 (post intervention period to assess rebound effect) [Note: a trend of change at each visit will also be assessed with respect to malaria seasonality]
Clinical malaria incidence from month 0 till months 12 and 20 of follow up | at months 0, 12 and 20
  number of symptomatic malaria episodes during and after intervention period

SECONDARY OUTCOMES:
Prevalence of asymptomatic malaria infections at month 0, 12 and 20 of follow up | from month 0 till month12 and 20
  to be measured from microscopic detection of malaria parasite on blood slides
Prevalence of PCR confirmed sub-microscopic parasitaemia at months 0,12 and 20 of follow up | at months 0, 12 and 20
  Polymerase chain reaction (PCR) confirmed from random subset of finger prick dry blood spots samples
Prevalence of soil transmitted helminths and schistosomiasis | at baseline, at month 12 and month 20.
  A stool sample will be used to determine prevalence (defined as adult or eggs) of STH and S. mansoni infection determined by duplicate Kato-Katz thick smears technique. Urine samples will be visually examined for the presence of blood (macrohaematuria) followed by laboratory examination for schistosomiasis infection (S.haematobium)
Prevalence of schistosomiasis | at baseline, at month 12 and month 20.
  Urine samples will be visually examined for the presence of blood (macrohaematuria) followed by laboratory examination for schistosomiasis infection (S.haematobium) for confirmation.
Prevalence of validated common P. falciparum polymorphisms known to be associated with drug sensitivity at baseline, at months 12 and 20 | at baseline, at month 12 and 20.
  from random subset of finger prick dry blood spots samples
Proportion of children seropositive for Plasmodium falciparum AMA-1 and MSP-119 at baseline, at month 12 and 20 | at baseline, at month 12 and 20.
  from random subset of finger prick dry blood spots samples, Antibody responses to P. falciparum blood-stages antigens, apical membrane antigen (AMA-1) and merozoite surface protein (MSP-119) will be determined.
Change in serum antibody responses to Plasmodium falciparum AMA-1 and MSP-119 at baseline, at month 12 and 20 | at baseline, at month 12 and 20.
  From random subset of finger prick dry blood spots samples to be eluted for ELISA
Percentages of school children with malnutrition through WHO's BMI z-score | at month 0, 12, and 20
  weight in kilograms and height in meters will be combined to report BMI in kg/m^2
Relative risk (RR), for all adverse events categorised to severity at month 12 and 20 | at month 12 and 20
  Adverse events will be detected throughout the study, Each intervention arm will be compared to control arm to determine risk of an adverse event among the two arms. Also events in two intervention arms will be compared to each other to assess risk in the two intervention arms.

OTHER OUTCOMES:
number of days missed school attendance pre and post intervention period | at baseline, at month 12 and 20
  number of days absent from school pre and post intervention period
Change in educational performance | at baseline, at month 12 and 20
  measured by annual change in average score of educational performance pre and post intervention period [to be provided by respective class teachers]
change in sustained attention on cognition evaluated using two code transmission tasks using TEA-Ch | evaluated at baseline, at month 12 and 20.
  sub group of 20 students selected at random in each class will be involved, sustained attention will be evaluated using two code transmission tasks, adapted from the Test of Everyday Attention for Children (TEA-Ch)
change in psychomotor functions tested by 20mShuttle Run Test pre and post intervention | evaluated at baseline, at month 12 and 20.
  sub group of 20 students selected at random in each class will be involved.Physical fitness will also be assessed using the 20 meter Shuttle Run Test (20mSRT). During this test children run continuously between two lines apart turning when signalled to do so by recorded beeps and a "shuttle" is defined as a run between one line to another. The 20mSRT has 20 levels.
Proportion of participants accepting IPTsc, using and completing dose of given study drugs. | at baseline, month 4, and 8
  This will be useful on future pragmatic implementation
Comparison of cost effectiveness of intervention between groups. | at month 12.
  Evaluated by assessing the implementation cost (setup, salaries, transport, price scenarios, etc), the study impact as well as possible synergies with other school health intervention programs. In addition,cost per child treated per year, the cost per anaemia case averted and cost per case P. falciparum parasitaemia averted as a result of the intervention, will also be evaluated to determine cost effectiveness of the program.

CONTACTS AND LOCATIONS:
Overall Officials: John PA Lusingu, MD, PhD, Principal Investigator — National Institute for Medical Research, Tanzania; Jean-pierre Van geertruyden, MD, PhD, Principal Investigator — Global health institute, University of Antwerp, Belgium.
Locations (1):
- National Institute for Medical Research, Tanga, Tanzania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hhera JJ, Makenga G, Baraka V, Francis F, Nakato S, Gesase S, Mtove G, Madebe R, Kyaruzi E, Minja DTR, Lusingu JPA, Van Geertruyden JP. Malaria-malnutrition interaction: prevalence, risk factors, and the impact of intermittent preventive therapy for malaria on nutritional status of school-age children in Muheza, Tanga, Tanzania - A cross-sectional survey and a randomized controlled open-label trial. BMC Public Health. 2025 Aug 13;25(1):2754. doi: 10.1186/s12889-025-23315-w. PMID 40804388
- [Derived] Makenga G, Baraka V, Francis F, Nakato S, Gesase S, Mtove G, Madebe R, Kyaruzi E, Minja DTR, Lusingu JPA, Geertruyden JV. Effectiveness and safety of intermittent preventive treatment with dihydroartemisinin-piperaquine or artesunate-amodiaquine for reducing malaria and related morbidities in schoolchildren in Tanzania: a randomised controlled trial. Lancet Glob Health. 2023 Aug;11(8):e1277-e1289. doi: 10.1016/S2214-109X(23)00204-8. PMID 37474234
- [Derived] Makenga G, Baraka V, Francis F, Nakato S, Gesase S, Mtove G, Madebe R, Kyaruzi E, Minja DTR, Lusingu JPA, Van Geertruyden JP. Effectiveness and safety of intermittent preventive treatment for malaria using either dihydroartemisinin-piperaquine or artesunate-amodiaquine in reducing malaria related morbidities and improving cognitive ability in school-aged children in Tanzania: A study protocol for a controlled randomised trial. Contemp Clin Trials Commun. 2020 Feb 20;17:100546. doi: 10.1016/j.conctc.2020.100546. eCollection 2020 Mar. PMID 32382685